CLINICAL TRIAL: NCT00067457
Title: A 12-Week, Randomized, Double-Blind, Placebo- Controlled Study of PRN BID and Fixed Dosing Regimens of Alosetron in Female Subjects With Severe Diarrhea-Predominant Irritable Bowel Syndrome Who Have Failed Conventional Therapy
Brief Title: Study In Women With Severe Diarrhea-Predominant Irritable Bowel Syndrome Having Failed Conventional Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S3B30048
Record Dates: First submitted 2003-08-20; First posted 2003-08-21 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Colon; Irritable Bowel Syndrome (IBS)
Keywords: PRN; Diarrhea-Predominant Irritable Bowel Syndrome; Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alosetron

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of as needed versus fixed dosing of an investigational medication for women with severe diarrhea-predominant Irritable Bowel Syndrome (IBS) who have failed conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe diarrhea-predominant Irritable Bowel Syndrome (IBS).
* Failed conventional therapy.
* Willing to make daily calls on a touch-tone telephone.

Exclusion criteria:

* History of or current chronic or severe constipation.
* Bloody diarrhea, abdominal pain with rectal bleeding.
* Thrombophlebitis.
* Abnormal thyroid stimulating hormone (TSH) value.
* Alcohol and/or substance abuse within past two years.
* Pregnant or lactating.
* History/treatment of malignancy within past five years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2003-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Subject self assessment of improvement between treatment groups using the IBS Global Improvement Scale; comparison of safety and tolerability between treatment groups with respect to adverse events & laboratory abnormalities. | 12 Weeks

SECONDARY OUTCOMES:
Comparison of treatment groups with respect to subject relief of IBS pain & discomfort; lower GI symptoms, changes in quality of life, lost workplace productivity, & lost household/leisure activity, & subject satisfaction with assigned study drug. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (170):
- United States (169):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Pell City, Alabama
  - GSK Investigational Site, Tallassee, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Carlsbad, California
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Bristol, Connecticut
  - GSK Investigational Site, Belleair Bluffs, Florida
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, Spring Hill, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Dunwoody, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Moline, Illinois
  - GSK Investigational Site, Morton Grove, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Clive, Iowa
  - GSK Investigational Site, Haysville, Kansas
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Florence, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Lanham, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Severna Park, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Northville, Michigan
  - GSK Investigational Site, Petoskey, Michigan
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Blackwood, New Jersey
  - GSK Investigational Site, Cedar Knolls, New Jersey
  - GSK Investigational Site, Oakhurst, New Jersey
  - GSK Investigational Site, Passaic, New Jersey
  - GSK Investigational Site, South Bound Brook, New Jersey
  - GSK Investigational Site, Willingboro, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Pittsford, New York
  - GSK Investigational Site, Pomona, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Jacksonville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bellbrook, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Wandsworth, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Levittown, Pennsylvania
  - GSK Investigational Site, Media, Pennsylvania
  - GSK Investigational Site, Morrisville, Pennsylvania
  - GSK Investigational Site, Penndel, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Stoneboro, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Conroe, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Pasadena, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Lacey, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
- GSK Investigational Site, Nedlands, Western Australia, Australia